CLINICAL TRIAL: NCT06240455
Title: A Double-blind, Placebo-controlled, Phase 2 Dose-range Study to Assess the Efficacy and Safety of WP1302 in Preventing Disease Relapse Following Methimazole Withdrawal in Subjects With Graves' Disease
Brief Title: Phase 2 Study to Assess Efficacy & Safety of WP1302 Prevent Relapse of MMI w/Draw in Subj. w/ Graves' dz
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Not feasible to recruit suitable subjects
Sponsor: Worg Biotherapeutics Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WP1302-CS-002
Record Dates: First submitted 2024-01-04; First posted 2024-02-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Graves Disease
Keywords: Graves' disease; preventing disease relapse; relapse rate; thyroid function
MeSH Terms: conditions — Graves Disease | interventions — Methimazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- WP1302 400μg (Active Comparator): After screening, eligible subjects will be randomized to treatment at a ratio (stratified by size of goiter [grade 0 or 1; grade 2], WHO classification) of 1:1:1:1 to either any group of MMI with WP1302 at a dose of 400 μg, 800 μg, or 1200 μg, or the group of MMI with placebo.
  The study consists of up to 5 periods: a screening period of up to 2 weeks; a WP1302 or placebo titration with MMI period of 12 weeks; a Full dose of WP1302 or placebo with MMI tapering period of 26 weeks; a follow-up period of 4 weeks; and an extended follow-up period of 6 months.
  Interventions: Drug: WP1302; Combination Product: methimazole
- WP1302 800μg (Active Comparator): After screening, eligible subjects will be randomized to treatment at a ratio (stratified by size of goiter [grade 0 or 1; grade 2], WHO classification) of 1:1:1:1 to either any group of MMI with WP1302 at a dose of 400 μg, 800 μg, or 1200 μg, or the group of MMI with placebo.
  The study consists of up to 5 periods: a screening period of up to 2 weeks; a WP1302 or placebo titration with MMI period of 12 weeks; a Full dose of WP1302 or placebo with MMI tapering period of 26 weeks; a follow-up period of 4 weeks; and an extended follow-up period of 6 months.
  Interventions: Drug: WP1302; Combination Product: methimazole
- WP1302 1200μg (Active Comparator): After screening, eligible subjects will be randomized to treatment at a ratio (stratified by size of goiter [grade 0 or 1; grade 2], WHO classification) of 1:1:1:1 to either any group of MMI with WP1302 at a dose of 400 μg, 800 μg, or 1200 μg, or the group of MMI with placebo.
  The study consists of up to 5 periods: a screening period of up to 2 weeks; a WP1302 or placebo titration with MMI period of 12 weeks; a Full dose of WP1302 or placebo with MMI tapering period of 26 weeks; a follow-up period of 4 weeks; and an extended follow-up period of 6 months.
  Interventions: Drug: WP1302; Combination Product: methimazole
- WP1302 Placebo (Placebo Comparator): After screening, eligible subjects will be randomized to treatment at a ratio (stratified by size of goiter [grade 0 or 1; grade 2], WHO classification) of 1:1:1:1 to either any group of MMI with WP1302 at a dose of 400 μg, 800 μg, or 1200 μg, or the group of MMI with placebo.
  The study consists of up to 5 periods: a screening period of up to 2 weeks; a WP1302 or placebo titration with MMI period of 12 weeks; a Full dose of WP1302 or placebo with MMI tapering period of 26 weeks; a follow-up period of 4 weeks; and an extended follow-up period of 6 months.
  Interventions: Drug: WP1302 placebo; Combination Product: methimazole

INTERVENTIONS:
Drug: WP1302 — Each arm will be treated with methimazole. During the MMI tapering period, commences the MMI weaning by reducing the original dosage by 50%. This adjusted dose is to be administered over a two-week duration. Continue this dose reduction in the subsequent 2-week durations until achieving a dose of 2.5 mg/day or lower. Upon reaching this threshold, MMI is to be discontinued (withdrawal).
  Arms: WP1302 1200μg; WP1302 400μg; WP1302 800μg
Drug: WP1302 placebo — Each arm will be treated with methimazole. During the MMI tapering period, commences the MMI weaning by reducing the original dosage by 50%. This adjusted dose is to be administered over a two-week duration. Continue this dose reduction in the subsequent 2-week durations until achieving a dose of 2.5 mg/day or lower. Upon reaching this threshold, MMI is to be discontinued (withdrawal).
  Arms: WP1302 Placebo
Combination Product: methimazole — Each arm will be treated with methimazole. During the MMI tapering period, commences the MMI weaning by reducing the original dosage by 50%. This adjusted dose is to be administered over a two-week duration. Continue this dose reduction in the subsequent 2-week durations until achieving a dose of 2.5 mg/day or lower. Upon reaching this threshold, MMI is to be discontinued (withdrawal).

SUMMARY:
This is a Phase 2, double-blind, placebo controlled, Methimazole (MMI) withdrawal study in subjects with Graves' disease. The study consists of up to 5 periods: a screening period of up to 2 weeks; a WP1302 or placebo titration with Methimazole period of 12 weeks; a Full dose of WP1302 or placebo with Methimazole tapering period of 26 weeks; a follow-up period of 4 weeks; and an extended follow-up period of 6 months.

After screening, eligible subjects will be randomized to treatment at a ratio (stratified by size of goiter [grade 0 or 1; grade 2], WHO classification) of 1:1:1:1 to either any group of Methimazole with WP1302 at a dose of 400 μg, 800 μg, or 1200 μg, or the group of Methimazole with placebo.

All the subjects will subsequently be enrolled in an extended safety follow-up period for an additional 6 months. Subjects who remain euthyroid will continue to be monitored for efficacy during the long-term follow-up.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, placebo controlled, Methimazole (MMI) withdrawal study in subjects with Graves' disease. The study consists of up to 5 periods: a screening period of up to 2 weeks; a WP1302 or placebo titration with Methimazole period of 12 weeks; a full dose of WP1302 or placebo with Methimazole tapering period of 26 weeks; a follow-up period of 4 weeks; and an extended follow-up period of 6 months.

After screening, eligible subjects will be randomized to treatment at a ratio (stratified by size of goiter [grade 0 or 1; grade 2], WHO classification) of 1:1:1:1 to either any group of Methimazole with WP1302 at a dose of 400 μg, 800 μg, or 1200 μg, or the group of Methimazole with placebo.

Subjects who have a confirmed diagnosis of Graves' disease based on medical history and/or physical examination and laboratory evidence, well controlled, with normalized thyroid function tests, and have received stable background Methimazole (i.e., not requiring dose adjustments) not exceeding 20 mg daily for at least 8 weeks and no more than 24 weeks are eligible to this study. All subjects enrolled in this study will receive Methimazole treatment in titration period.

During the titration period, subjects will receive WP1302 or placebo by subcutaneous (S.C.) injection every 2 weeks (Q2W) for 12 weeks while continuing MMI (see "Dosing" below). The dose of WP1302 will be titrated up to the target dose assigned to the subject during this period (see "Dosing" below). Thyroid symptoms and function tests will be evaluated every 2 weeks. The investigator may adjust the frequency of thyroid function tests based on safety considerations. If a subject does not maintain euthyroidism, which is defined as total T3 60-180 ng/dL, free T4 0.8-1.8 ng/dL, and TSH 0.5-5 mU/L, during the "WP1302 titration period", the subject will be discontinued from Investigational Medicinal Product (IMP) (i.e., WP1302 or placebo) and the subject is still required to complete the end-of study visit.

During the 26-week full dose of WP1302 with Methimazole tapering period, subjects who have maintained euthyroidism during the "WP1302 titration period" will be dosed with WP1302 at 400, 800, or 1200 μg with down-titrated Methimazole. Thyroid symptoms and function tests will be evaluated every 2 weeks. The investigator may adjust the frequency of thyroid function tests based on safety considerations. Subjects who experience disease relapse will be treated with Methimazole as first-line therapy (see "Management of Relapse and Rescue Medication" below).

At the end of the full dose of WP1302 with Methimazole tapering period, subjects will have 4 weeks of follow-up, and complete an end-of-study visit at Week 42. All the subjects will subsequently be enrolled in an extended safety follow-up period for an additional 6 months. Subjects who remain euthyroid will continue to be monitored for efficacy during the long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years at the time of informed consent.
2. Confirmed diagnosis of Graves' disease through medical history and/or physical examination, laboratory evidence as documented by a serum TSH<0.5 mU/L and either a serum total T3 >180 ng/dL or a serum free T4 > 1.8 ng/dL.
3. Current use of MMI at stable dose not exceeding 20 mg daily for at least 8 weeks and no more than 24 weeks by the baseline (Week 0).
4. 60 ng/dL < serum total T3 ≤ 180 ng/dL, 0.8 ng/dL < serum free T4 ≤1.8 ng/dL, and 0.5 mU/L ≤ serum TSH <5 mU/L at the Screening Visit.
5. Willing and able to give written informed consent, agree to provide contact with the endocrinologist (or other appropriate trained healthcare provider), and to comply with protocol assessments/procedures.
6. Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study, and until at least 6 months after the last dose of WP1302.

Female subjects of child-bearing potential must use a highly effective method of contraception throughout the entire duration of the study and for at least 6 months after the last dose of WP1302.

Exclusion Criteria:

1. Currently using biotin supplements.
2. Known history of allergy to the ingredients of WP1302, or hypersensitivity reaction that in the opinion of the investigator would exclude the subject's participation in the study.
3. Previous treatment with radioiodine or (partial or complete) thyroidectomy.
4. Subjects with known pituitary disease, such as traumatic brain disease, hyperprolactinemia, and hypophysitis.
5. Treatment with steroids (administered via the oral and/or parenteral routes) within 3 months prior to baseline or requiring intermittent use of systemic steroids for disease management (such as severe asthma), inhaled steroids are not prohibited.
6. History of hyperthyroidism not caused by Graves' disease (e.g., toxic multinodular goiter, autonomous thyroid nodule, or acute inflammatory thyroiditis).
7. Subjects who may have thyroid nodules that require alternative intervention.
8. Symptoms and signs of thyroid storm such as fever, profuse sweating, vomiting, diarrhea, delirium, severe weakness, seizures, markedly irregular heartbeat, yellow skin and eyes (jaundice), severe low blood pressure, and coma, pyrexia with no other cause than hyperthyroidism.
9. Subjects who have a history of intolerance or contraindication to the use of beta-blockers.
10. Subjects with history of arrhythmia, or cardiovascular accident, or other cardiovascular disease who maybe at increased risk of cardiac adverse events from treatment or recurrence of hyperthyroidism.
11. Subjects with history of cerebrovascular accident/transient ischemic attack, or other cerebrovascular disease who maybe at increased risk of neurologic adverse events from treatment or recurrence of hyperthyroidism.
12. Prior treatment with immunotherapies (including rituximab), any cytokine or anti-cytokine therapy.
13. Prior treatment with immunomodulatory drugs, such as cyclosporine A, methotrexate, and/or cyclophosphamide.
14. Prior use of disease-related T cell-inducing therapy or peptide-tolerizing agent to treat Graves' disease.
15. Inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase > 3 times the upper limits of the normal (ULN) at screening.
16. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2, calculated as individual eGFR derived from Modification of Diet in Renal Disease formula.
17. Receiving hemodialysis or peritoneal dialysis or microdialysis or continuous venovenous hemofiltration or continuous venovenous hemodialysis.
18. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
19. Known history of active or chronic infectious disease or any disease which compromises immune function (e.g., HIV+, HTLV-1, active Lyme disease, latent or active TB, viral hepatitis).
20. Major surgery within 6 months prior to the screening visit or requiring ongoing active treatment after surgery irrespective of the time since surgery.
21. Active thyroid eye disease (clinical activity score [CAS] ≥3) with functional visual impairment sufficient to cause poor quality of life, or dysthyroid optic neuropathy likely to require immunosuppressive treatment during the 30 weeks of the study.
22. Any vaccination within 30 days prior to screening, except for influenza and coronavirus vaccines.
23. Being pregnant, breastfeeding, or planning to become pregnant during the study.
24. Documented presence of immunodeficiency or an immunocompromised condition including hematologic malignancy, bone marrow transplant, or known human immunodeficiency virus infection with a CD4 count <200/mm3.
25. Currently actively moderate-heavy using tobacco (≥10 cigarettes a day).
26. Participating in any clinical study of any investigational medication (i.e., unauthorized medication) within 90 days prior to randomization.
27. Any other significant medical illness or psychiatric conditions that in the opinion of the investigator, would preclude participation in the study or impair the ability to give informed consent; any other clinically apparent autoimmune disease currently requiring disease-modifying or anti-inflammatory treatment; or significant illness which has not resolved within 4 weeks prior to the planned date of first dose of WP1302.
28. Any other conditions or prior therapies, which, in the opinion of the investigator, would make the subject unsuitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | Up to 42 weeks
  To assess the relapse rate between the WP1302 and placebo treatment groups in subjects who enter the tapering phase

SECONDARY OUTCOMES:
Replase time | Up to 42 weeks
  To assess the time duration from start of methimazole (MMI) tapering to disease relapse between the subjects treated with WP1302 and placebo.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 68 weeks including LTFU
  To assess the safety and tolerability of WP1302 administered with or without methimazole (MMI) in subjects with Graves' disease
Total T3, free T4, and TSH levels | Up to 68 weeks including LTFU
  To assess the effect of WP1302 on thyroid function (measured by total T3, free T4, and TSH levels)
Pharmacokinetics (PK) parameters (AUC, Cmax) | Week 0 and Week 10
  To assess the pharmacokinetics (PK) parameters (AUC, Cmax) of WP1302 in plasma
Incidence of anti-drug antibodies (ADAs) | Up to 68 weeks including LTFU
  To assess the incidence of anti-drug antibodies (ADAs) against WP1302

OTHER OUTCOMES:
Cytokine levels of IFN-γ, IL-2, IL-6, and IL-10 | Up to 42 weeks
  To assess the effects of WP1302 on immune response by measuring the plasma cytokine levels of IFN-γ, IL-2, IL-6, and IL-10
TSH receptor antibody (TRAb) levels | Up to 68 weeks including LTFU
  To assess the effects of WP1302 on TSH receptor antibody (TRAb)
HLA haplotypes | Baseline
  To assess potential correlations between response to WP1302 and HLA haplotypes
Thyroid eye disease (TED) condition | Up to 42 weeks
  To assess occurrence, severity, and changes in severity of thyroid eye disease (TED) in a subset of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Lee, MD, Study Chair — Worg Biotherapeutics Inc.
Locations (7):
- United States (7):
  - East Valley Diabetes and Endocrinology-Clinical Research, PLLC, Hunt, Arizona
  - Alliance Research Institute, Canoga Park, California
  - Paradigm Clinical Research Centers - Littleton, Littleton, Colorado
  - BayCare Health System, Inc., Clearwater, Florida
  - Albuquerque Clinical Trials Inc, Albuquerque, New Mexico
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Research Solution LLC dba Endocrine and Psychiatry Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No